CLINICAL TRIAL: NCT04660500
Title: Driving Performance of People With Parkinson's Using Autonomous In-Vehicle Technologies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Disability, Independent Living, and Rehabilitation Research (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB202002321; 90IFRE0035-03-00 (Other Grant/Funding Number: ADMIN FOR COMMUNITY LIVING)
Record Dates: First submitted 2020-11-30; First posted 2020-12-09 (Actual); Last update posted 2024-01-19 (Actual); Status verified 2024-01

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; In-vehicle information system; Advanced driver assistance system
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PD Drivers Using AV Technologies On-road (Experimental): Each driver will drive on-road, everybody will be exposed to two drives (Drive 1, Drive 2) one drive with and the other without in-vehicle technology. The order of technology (with vs. without IVIS or ADAS) and the order of the routes (Drive 1 vs. Drive 2) will be randomly allocated to control for order effects.
  Interventions: Other: PD Drivers Using AV Technologies On-road

INTERVENTIONS:
Other: PD Drivers Using AV Technologies On-road — All drives will include events to assess the impact of in-vehicle information systems (IVIS) and advanced driver assistance systems (ADAS) on the driving performance (driving errors) of drivers with PD. For IVIS the investigators will include options to assess errors with lane maintenance (with and without the lane departure warning system) and signaling (with and without blind spot detection). For ADAS the investigators will include conditions to assess errors in speeding (with and without adaptive cruise control) and lane exceedances (with and without lane keeping assist).

SUMMARY:
For drivers with Parkinson's Disease (PD), autonomous in-vehicle technologies may help mitigate functional deficits, improve driving performance, decrease driving errors and enhance their ability to stay on the road. Using a pretest/posttest design the investigators will quantify the use of In-vehicle Information Systems (IVIS) and Advanced Driver Assistance Systems (ADAS) during driving to illustrate how IVIS and ADAS may affect driving, and provide recommendations to drivers with PD, the clinical community and industry.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects diagnosed by a neurologist/ movement disorder specialist with clinically probable PD by Movement Disorders Society (MDS) criteria 25
2. Has mild or moderate disease severity, based on the MDS-Unified Parkinson's Disease Rating Scale for motor symptoms (hereafter referred to as the UPDRS section 3) in the on state of medications (i.e., one hour of taking PD medications) and the Modified Hoehn and Yahr disease severity scale
3. Is representative of one of two PD groups based on age, i.e., participants with symptom onset between 35-64 years of age (younger onset), or participants with symptom onset between ages 65- 85 years (older onset)
4. Currently driving with a valid license
5. Meets the Florida state requirement for visual acuity of at least 20/50 in one eye, if one eye is blind or 20/200 or worse the other eye must be 20/40 or better (20/40 in at least one eye) and field of vision (130 degrees or more)
6. Lives independently in the community
7. Proficient in reading/speaking English
8. A Montreal Cognitive Assessment (MoCA) score of 20 or higher

Exclusion Criteria:

1. Concurrent neurological conditions (e.g., stroke, seizures; dementia)
2. Severe psychiatric (e.g., psychoses/ significant anxiety) or physical conditions (e.g., missing limbs) precluding full participation
3. Use of psychotropic medications having adverse effect on mental/physical functioning
4. Severe, unpredictable motor fluctuations
5. Severe sleep difficulties.

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Total number of driving errors | 1 year up to study completion
  The evaluator will record the total number of driving errors by number and type (i.e., speeding, lane maintenance, and signaling) on a standardized data collection form.
Type and number of driving errors | 1 year up to study completion
  Type of driving errors include: speeding, lane maintenance and signaling on-road recorded by the evaluator, or via vehicle recorded kinematics and telematics (e.g., in-vehicle GPS to record speed).

CONTACTS AND LOCATIONS:
Overall Officials: Sherrilene Classen, PhD, Principal Investigator — University of Florida
Locations (1):
- UF Norman Fixel Institute for Neurological Diseases, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Classen S, Li Y, Giang W, Winter S, Wei J, Patel B, Jeghers M, Gibson B, Rogers J, Ramirez-Zamora A. RCT protocol for driving performance in people with Parkinson's using autonomous in-vehicle technologies. Contemp Clin Trials Commun. 2022 Jun 28;28:100954. doi: 10.1016/j.conctc.2022.100954. eCollection 2022 Aug. PMID 35812823